## **INFORMED CONSENT**

NCT05825755

2024/01/04

## **Participant Consent**

| Research title: |
|---|
| "Randomized multicenter study for the validation of the HumanITcare platform." Protocol code: FOLLOWHEALTH-2023-02 (Version 2, 06/13/2023). Center: |
| They, |
| // <del></del> |
| - I have read the information sheet that has been given to me about the |
| investigation I have been able to ask questions about the investigation. |
| - I have received sufficient information about the investigation. |
| - I have spoken with: (name of researcher) |
| - I understand that my participation is voluntary. |
| - I understand that I can withdraw from the research: |
| - Whenever you want. |
| - Without having to give explanations. |
| - Without this affecting my medical care. |
| and of the Council of April 26, 2016 regarding the protection of natural persons with regard to the processing of personal data and the free circulation of data, I declare that I have been informed of the existence of a file or processing of personal data, the purpose of its collection and the recipients of the information. - I freely give my consent to participate in the research. Signature of |
| participant Signature of researcher |
| Date:/ Date:/ |
| I want you to communicate to me the information derived from the research that may be relevant to my health: |
| □ AND □ NO |
| Signature of Participant Signature of Investigator Date:/ Date: |

## **Revocation of consent:**

| The und | lersign | ed pat | ient revoke | es the o | consent granted to the doctor Dr. |
|---|---|---|---|---|---|
| | | | | | for his participation in the "Randomize |
| multicer | nter st | udy fo | r the valida | ition of | the HumanITcare platform." |
| Doublein | م ماام د | : | ua Dhuaisia | nla Ciau | |
| Participa | ant S S | ignatu | re Physicia | n s Sigi | lature |
| Date: | / | / | Date: | / | / |